CLINICAL TRIAL: NCT03167554
Title: Effectiveness of Therapeutic Percutaneous (EPTE®) Guided by Ultrasound as a Treatment of Achilles Tendinopathy. A Randomized Controlled Clinical Trial.
Brief Title: Ultrasound Guided Therapeutic Percutaneous Electrolysis in Achilles Tendinopathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HUILeonor
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Electrolysis; Achilles Tendinopathy; Ultrasonography; Physical Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham group (Sham Comparator): Simulating of the electrolysis application.he electrolysis technique was simulated to be delivered. The guide tube of the needle contacted with the skin, located on the painful area, and the device remained switched on to simulate its functioning.
  Interventions: Other: Sham comparator
- Experimental group 1 (Experimental): Electrolysis application with monopolar needle.
  Interventions: Other: Experimental group 1
- Experimental group 2 (Experimental): Electrolysis application with bipolar needle.
  Interventions: Other: Experimental group 2

INTERVENTIONS:
Other: Sham comparator — The electrolysis technique was simulated to be delivered. The guide tube of the needle contacted with the skin, located on the painful area, and the device remained switched on to simulate its functioning.
  Other Names: Sham group
  Arms: Sham group
Other: Experimental group 1 — Percutaneous Therapeutic Electrolysis (EPTE®) with monopolar needle, 330 microamps, 1 min 20 sec.
  Other Names: Electrolysis application with monopolar needle.
  Arms: Experimental group 1
Other: Experimental group 2 — Percutaneous Therapeutic Electrolysis (EPTE®) with bipolar needle, 120 microamps, 1 min 20 sec.
  Other Names: Electrolysis application with bipolar needle.
  Arms: Experimental group 2

SUMMARY:
Achilles tendon is a frequent lower-limb tissue where tendinopathy may arise. Percutaneous Therapeutic Electrolysis (EPTE®) is an electronic device that enables to treat accurately, guided by an ultrasound, the tendon injured area by applying a galvanic current through an acupuncture needle. Thus, the first stage of physiological regenerative process may be obtained. Design: Randomized Controlled Clinical Trial. Objectives: To know the effectiveness of Percutaneous Therapeutic Electrolysis (EPTE®) versus a sham intervention at improving pain and function in patients who undergo Achilles Chronic Tendinopathy and to determine the efficiency of Percutaneous Therapeutic Electrolysis (EPTE®) with monopolar needle versus Percutaneous Therapeutic Electrolysis (EPTE®) with bipolar needle at improving pain and function in patients who undergo Achilles Chronic Tendinopathy. Participants: patients diagnosed with Achilles Chronic Tendinopathy. Setting. Infanta Leonor Hospital, Madrid, Spain. Experimental intervention: Percutaneous Therapeutic Electrolysis (EPTE®) with monopolar needle, 330 microamps, 1 min 20 sec versus bipolar needle. Sham intervention: the guide tube of the needle contacted with the skin and the device remained switched on to simulate its functioning.

DETAILED DESCRIPTION:
Tendinopathy is a common injury among athletes, where the incidence reaches 50%. Nevertheless, industrial workers as well as sedentary subjects may also undergo this pain condition.

Achilles tendon is a frequent lower-limb tissue where tendinopathy may arise. Achilles tendinopathy risk factors have been detailed, such as: age, mechanical axis deviation of lower limbs, excessive training load dosage, and type of work activity. The middle portion of the tendon is the area where Achilles tendinopathy is most likely to be located. Interestingly, correlation between pain severity and the degree of tissue degeneration by imaging diagnosis is hardly showed in chronic tendinopathy conditions. Thus, chronic tendinopathy pain may be mediated not only by peripheral but by central mechanisms.

Percutaneous Therapeutic Electrolysis (EPTE® System; Manual EPTE, 2014 IONCLINICS & DEIONIC, S.L.) is an electronic device that enables to treat accurately, guided by an ultrasound, the tendon injured area by penetrating the skin with an acupuncture needle. A galvanic current goes through the device to the needle so that the first stage of physiological regenerative process may be obtained. That is due to a chemical reaction that leads to a controlled alkaline burn into the injured tissue and a subsequent basification of extracellular medium. That elicits an inflammatory response; the destroyed tissue is metabolized by phagocytosis process. Design: Randomized Controlled Clinical Trial. Objectives: To know the effectiveness of Percutaneous Therapeutic Electrolysis (EPTE®) versus a sham intervention at improving pain and function in patients who undergo Achilles Chronic Tendinopathy, and to determine the efficiency of Percutaneous Therapeutic Electrolysis (EPTE®) with monopolar needle versus Percutaneous Therapeutic Electrolysis (EPTE®) with bipolar needle at improving pain and function in patients who undergo Achilles Chronic Tendinopathy. Participants: patients diagnosed with Achilles Chronic Tendinopathy. Setting. Infanta Leonor Hospital, Madrid, Spain. Experimental intervention: Percutaneous Therapeutic Electrolysis (EPTE®) with monopolar needle, 330 microamps, 1 min 20 sec versus bipolar needle. Sham intervention: the guide tube of the needle contacted with the skin and the electrolysis device remained switched on to simulate its functioning.

ELIGIBILITY:
Inclusion Criteria:

- Achilles Chronic Tendinopathy diagnosis (from 3months up to 3 years)

Exclusion Criteria:

* Physical therapy treatment within the last 4 months.
* Surgery approach for Achilles tendinopathy.
* Pregnancy
* Corticoid treatment in the last 4 months.
* Pacemaker
* Thrombophlebitis
* Systemic disease
* Cognitive disease
* Prosthesis or osteosynthesis
* Dermatopathies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 5 min
  Measured by Numeric Pain Rating Scale. Punctuation from 0 point up to 10 points. "0" no pain; "10" the most bearable pain.

SECONDARY OUTCOMES:
Lower limb functionality | 10 min
  Measured by Visa-A Scale. Punctuation from 0 point up to 100 points. "0"point the most inability; "100" points complete functionality.
Achilles tendon thickening | 5 min
  Assessed by ultrasonography. Thickening was considered when the thickness is 50% greater than the contralateral limb.
Length of the most thickened area | 5 min
  Assessed by ultrasonography. Distance (in mm) between the two extremes of the thickened area
Location of the most thickened area | 5 min
  Assessed by ultrasonography. Distance (in mm) from the Achilles insertion up to the thickening onset.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Herraiz Garvin, MSc, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (1):
- Hospital Universitario Inflanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided